CLINICAL TRIAL: NCT06657391
Title: Evaluation of the Clinical Efficacy and Safety of Recombinant Humanized Anti-CD25 Monoclonal Antibody in Preventing Graft-versus-host Disease After Haploidentical / Matched Unrelated Donor Hematopoietic Stem Cell Transplantation in Patients with Transfusion-dependent Thalassemia: a Prospective, Multicenter, Open-label, Randomized Controlled Clinical Trial
Brief Title: Evaluation of Recombinant Humanized Anti-CD25 Monoclonal Antibody for Preventing Graft-versus-host Disease After Haploidentical/matched Unrelated Donor Hematopoietic Stem Cell Transplantation in Patients with Transfusion-dependent Thalassemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rongrong Liu (Other)
Responsible Party: Sponsor-Investigator, Rongrong Liu, consultant; professor, First Affiliated Hospital of Guangxi Medical University
Organization: First Affiliated Hospital of Guangxi Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-K387-01
Record Dates: First submitted 2024-10-21; First posted 2024-10-24 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Transfusion Dependent Thalassemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The researchers and the subjects wil aware of the grouping and the intervention they received. However, this trail will implement a blind method for the outcomes assessors, who objectively evaluated the outcome indicators without knowing the grouping of the subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): The intervention group will receive 4 doses of recombinant humanized anti-CD25 monoclonal antibody (Sunshine Guojian Pharmaceutical(Shanghai) Co.,Ltd.) on days +7, +14, +28, and +42 after transplantation, with a recommended dose of 1 mg/kg.
  Interventions: Drug: recombinant humanized anti-CD25 monoclonal antibody
- control group (No Intervention): The control group will receive no treatment at the same time points.

INTERVENTIONS:
Drug: recombinant humanized anti-CD25 monoclonal antibody — The intervention group received 4 doses of recombinant humanized anti-CD25 monoclonal antibody on days +7, +14, +28, and +42 after transplantation, with a recommended dose of 1 mg/kg.
  Arms: intervention group

SUMMARY:
Graft-versus-host disease (GVHD) is a major factor affecting the efficacy and quality of life of alternative donor transplantation in thalassemia major (TM), severely limiting the clinical application of alternative donor transplantation in TM.The purpose of this clinical trial is to evaluate whether recombinant humanized anti-CD25 monoclonal antibody is effective in preventing GVHD and its safety after haploidentical/matched unrelated donor hematopoietic stem cell transplantation. The main questions it aims to answer are:

* Does recombinant humanized anti-CD25 monoclonal antibody reduce the incidence of GVHD disease after haploidentical/matched unrelated donor hematopoietic stem cell transplantation?
* What medical problems will participants experience when using the recombinant humanized anti-CD25 monoclonal antibody? What is the quality of life after 2 years follow-up? In this clinical trail, participants will be randomly assigned to the intervention group or the control group by researchers in a 2:1 ratio. The intervention group will be given recombinant humanized anti-CD25 monoclonal antibody (1mg/Kg) combined with the standard GVHD prophylaxis after transplantation, while the control group will only receive the standard GVHD prophylaxis. The incidence of GVHD after transplantation in the two groups will be observed. The main evaluation is the clinical efficacy of recombinant humanized anti-CD25 monoclonal antibody in preventing aGVHD.

ELIGIBILITY:
Inclusion Criteria:

* patients with transfusion-dependent thalassemia;
* patients who are planning to receive matched unrelated donor hematopoietic stem cell transplantation (MUD-HSCT) or HLA haploidentical donor hematopoietic stem cell transplantation (HID-HSCT);
* physical condition score (Lansky/Karnofsky score) ≥ 70%;
* patients (or legal guardians) voluntarily participate in the study and sign the informed consent form

Exclusion Criteria:

* patients with HLA-matched hematopoietic stem cell donors and willing to receive HLA-matched hematopoietic stem cell transplantation;
* patients with known infectious diseases such as hepatitis B, hepatitis C, AIDS, syphilis, human T-lymphotropic virus, etc.;
* patients with serious active bacterial, viral, fungal, malaria or parasitic infections;
* patients with autoimmune deficiency diseases;
* patients with a history of malignant tumors or current malignant tumors;
* patients with important organ diseases or abnormal laboratory tests, including but not limited to: 1) patients with cirrhosis, liver fibrosis or active hepatitis, and/or abnormal liver function tests (alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≥2.5×ULN; alkaline phosphatase ≥2.5×ULN); 2) patients with heart disease, or left ventricular ejection fraction (LVEF) <60%, or severe iron deposition in the heart; 3) kidney disease, or blood creatinine ≥1.5×ULN with creatinine clearance <30% of normal level; 4) patients with endocrine dysfunction;
* patients with uncorrected bleeding disease;
* patients with severe mental illness (such as severe depression, schizophrenia, etc.) or cognitive dysfunction (dementia, delirium, etc.), which are unable to cooperate with the study;
* peripheral blood white blood cell (WBC) count <3×10^9/L or platelet count <100×10^9/L;
* patients having received thalidomide treatment within the past 3 months;
* patients having received any type of gene and/or cell therapy in the past;
* patients with severe allergies;
* female patients who are pregnant, breastfeeding, or planning to become pregnant within 1 year of participating in this trial;
* patients who are participating in other clinical trials;
* other situations that are not suitable for participation in this clinical trial as assessed by the investigator.

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 396 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Grade III-IV aGVHD | within 100 days after HID-HSCT/MUD-HSCT
  the incidence of grade III-IV aGVHD within 100 days after HID-HSCT/MUD-HSCT was compared between the intervention group and the control group.

SECONDARY OUTCOMES:
Grade II-IV aGVHD | within 100 days after HID-HSCT/MUD-HSCT
  the incidence of grade II-IV aGVHD within 100 days after HID-HSCT/MUD-HSCT was compared between the intervention group and the control group.
Chronic graft-versus-host disease (cGVHD) | 2 years
  The incidence of cGVHD after HID-HSCT/MUD-HSCT was compared between the intervention group and the control group.
Overall survival (OS) | 2 years
  Comparison of 2-year OS between the intervention group and the control group.
Thalassemia-free survival (TFS) | 2 years
  comparison of the 2-year TFS between the intervention group and the control group.
Transplantation-related mortality (TRM) | 2 years
  comparison of the 2-year TRM between the intervention group and the control group.
Transplantation-related complications | 2 years
  comparison of the 2-year transplantation-related complications between the intervention group and the control group.
Infection | 2 years
  comparison of the infection during the transplantation between the intervention group and the control group.
Immune reconstitution | 2 years
  comparison of the immune reconstitution after transplantation between the intervention group and the control group.
Quality of life | 2 years
  comparison of the quality of life between the intervention group and the control group by using the Pediatric Quality of Life Inventory Version 4.0 (PedsQL4.0) scale. The scales are comprissed of parallel self-report and parent proxy-report formats:
  1. Self-report includes ages 8 to 12, 13 to 18, and 18 to 25, with a total of 23 items.
  2. Parent proxy-report assesses parent's perceptions of their child's health-related quality of life. Parent proxy-report (ages 5 to 7) has 23 items, and Parent proxy-report (ages 2 to 4) has 21 items.
  A 5-point response scale is utilized across self-report for ages and parent proxy-report (0 = never a problem; 1 = almost never a problem; 2 = sometimes a problem; 3 = often a problem; 4 = almost always a problem). Items are reverse-scored and linearly transformed to a 0 to 100 scale (0 = 100, 1 = 75, 2 = 50, 3 =25, 4 = 0), so that higher scores indicate better health-related quality of life.
Adverse events | 2 years
  comparison of the occurrence of adverse events between the intervention group and the control group.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Maoming People's Hospital, Maoming, Guangdong
  - Liuzhou Workers' Hospital, Liuchow, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Yulin Red Cross Hospital, Yulin, Guangxi
  - Hainan Provincial People's Hospital, Haikou, Hainan

IPD SHARING:
Plan to Share IPD: No